CLINICAL TRIAL: NCT05986084
Title: Linking HIV Prevention and Postpartum Care: Safety, Efficacy and Feasibility of Cabotegravir-LA PrEP in a High-Risk Breastfeeding Population in Botswana
Brief Title: Tshireletso: Safety, Efficacy and Feasibility of Cabotegravir-LA PrEP in a Breastfeeding Population in Botswana
Acronym: Tshireletso
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Botswana Harvard AIDS Institute Partnership (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Rebecca Zash, MD, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023P000415; 5R01HD108047 (NIH)
Record Dates: First submitted 2023-07-27; First posted 2023-08-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Pre-Exposure Prophylaxis (PrEP); Breast Feeding
Keywords: Botswana; Lactation; Infant PK; long acting injectable; HIV prevention; post-partum; integrase strand transfer inhibitor; cabotegravir
MeSH Terms: conditions — Breast Feeding | interventions — cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAB-LA PrEP (Experimental): Following a negative HIV test, long-acting Cabotegravir Injection (CAB-LA) 600mg will be administered as a 3mL intramuscular (IM) injection in the gluteal muscle at enrollment, 1 month, and then every 2 months, for a maximum of 13 injections over 24 months of follow up.
  Interventions: Drug: Cabotegravir Injection [Apretude]

INTERVENTIONS:
Drug: Cabotegravir Injection [Apretude] — Injection

SUMMARY:
The goal of this this hybrid safety/implementation study is to evaluate whether using long-acting cabotegravir (CAB-LA) for HIV prevention (PrEP) is acceptable, feasible and safe in post-partum people who are breastfeeding. The main question[s] it aims to answer are:

* Will CAB-LA injections work well as a way to prevent HIV infection in post-partum people?
* Will CAB-LA injections be safe in post-partum people and their infants who will be breastfeeding?

Participants without HIV who are admitted to the maternity ward after having delivered a baby will be offered to start CAB-LA PrEP. Those who choose to participate will receive their first dose (injection) at the maternity ward and their follow up doses (injections) at their local clinic when they come for routine post-partum and pediatric care. Participants and their infants will be followed in the study for 24 months. We will be following how many people come on-time for their CAB-LA injections, how often they keep coming back, and the reasons they continue (or stop) these injections. We will also test people for HIV at all of their visits to see how many people get HIV during the study. We will also measure the levels of the medication in the blood of the post-partum people and their infants (who may be getting some of the CAB-LA in breastmilk) and evaluate to see if their is any impact of CAB-LA on the health of the post-partum person or their infants.

DETAILED DESCRIPTION:
This is a hybrid implementation/safety study of long-acting cabotegravir (CAB-LA) as pre-exposure prophylaxis (PrEP) to prevent HIV infection in a post-partum cohort in Botswana where breastfeeding is common. The investigators will enroll 500 women at risk for HIV while they are admitted to the postpartum maternity ward after delivery at government-run health care facilities in Botswana and follow them for 24 months. The study sites will be located in two districts in Botswana, Gaborone and Molepolole.

The first CAB-LA injection will occur generally before discharge from the maternity ward. Follow up injections at 1 month, and then every 2 months, will be administered at clinics where the women and their infants receive routine care (or at research study sites when needed). The investigators will will measure uptake, adherence, persistence and implementation metrics using a mixed methods approach. The investigators will evaluate factors associated with uptake, adherence and persistence using data collected on all participants via questionnaires. The investigators will also conduct in-depth interviews of eligible participants who do not want CAB-LA and also a subset of enrolled participants at enrollment, 7 months and 19 moths. At each visit The investigators will screen for HIV using 4th generation HIV ag/ab point-of care tests and report HIV incidence over 24 months. The investigators will also evaluate safety outcomes, including postpartum depression, weight gain, and infant growth and INSTI resistance in incident HIV infections. Pharmacokinetics of CAB-LA in lactation (women, infants and breastmilk) will be evaluated in 30 mother-infant pairs in a PK substudy. HIV incidence and safety outcomes will be compared with a similar cohort of participants enrolled in a separate observational study in Botswana. This separate study also enrolls at the time of delivery from the same maternity sites.

ELIGIBILITY:
Inclusion Criteria:

1. Mother 18 years of age or older and willing and able to provide an informed consent
2. < 14 days after delivery (calendar day of birth = day 0)
3. Negative HIV screening test (conducted at the time of enrollment)
4. Mother <30 years old or has had < 3 prior pregnancies (Gravida 1, 2, or 3 including this pregnancy)
5. Plan to stay and receive postpartum and pediatric care in the Gaborone or Molepolole region for 24 months

Exclusion Criteria:

1. Receiving carbemazapine, phenobarbital, phenytoin, oxycarbazepine, rifampin, rifabutin, rifapentine, systemic dexamethasone (>1 dose oral/IV), or St. John's wort
2. Suspected to have, recently diagnosed with, or on treatment for TB (due to interaction with rifampin)
3. Previous hypersensitivity reaction to CAB or other INSTI
4. Unstable medical or psychiatric condition making it unlikely they will be able to adhere to injections every 8 weeks
5. Plan for pediatric and post-partum care outside the government system (private clinics)
6. Inflammatory skin condition that compromises the safety of the intramuscular injection
7. Weight <35kg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Persistence of CAB-LA injections | 24 months
  The % of participants continuing CAB-LA PrEP at 5 months,11 months,17 months and 24 months
Uptake of CAB-LA injections | 24 months
  The % of eligible participants accepting CAB-LA PrEP
Adherence to CAB-LA injections | 24 months
  The % of injection visits attended by participants
HIV Incidence | 24 months
  The incidence of HIV infections will be calculated as the number of HIV infections infections identified during follow up, per person-year)
Composite Maternal Adverse Effects | 24 months
  The % of participants with any of the following: grade 2 or higher DAIDS-graded adverse event, obesity (24 month BMI >30), new onset diabetes and pre-diabetes (HgBA1c >5.8 or diagnosis during routine care), hypertension (systolic >140 or diastolic >90 on 2 separate measurements, or diagnosis during routine care) and prevalence of depression (PHQ-9 score >9) or diagnosis during routine care
Composite Infant Adverse Effects | 24 months
  The % of infants with any of the following: incident pediatric HIV infections, Z-score >=2 standard deviations (SD) below norms for length-for-age, weight-for-age or head-circumference-for-age based on WHO growth curves at 24 months

SECONDARY OUTCOMES:
Maternal Cabotegravir Levels | 5 months
  Paired serum and breastmilk cabotegravir levels will be assessed just before the 1-month CAB-LA injection (early trough), 1 week after the 1-month CAB-LA injection (early peak), just before the 5-month CAB-LA injection (steady state trough) and 1 week after the 5-month CAB-LA injection (steady state peak)
Infant Cabotegravir Levels | 5 months
  In breastfed infants, infant serum cabotegravir levels will be assessed just before the 1-month CAB-LA injection (early trough), 1 week after the 1-month CAB-LA injection (early peak), just before the 5-month CAB-LA injection (steady state trough) and 1 week after the 5-month CAB-LA injection (steady state peak)
Median maternal weight change | 24 months
  The investigators will describe the median change in weight over the follow up period and the median weight gain from pre-pregnancy weight (when available)
Maternal Obesity | 24 months
  BMI >30 at 24 months
Maternal Diabetes | 24 months
  New onset diabetes and pre-diabetes (HgBA1c >5.8 or diagnosis during routine care)
Maternal Hypertension | 24 months
  Systolic blood pressure >140 and/or diastolic blood pressure >90 on 2 separate measurements, or diagnosis during routine care
Maternal Depression | 24 months
  PHQ-9 score >9 or diagnosis of post partum depression in routine care
Infant HIV infection | 24 months
  The % of infants diagnosed with HIV infection, per person-years of follow up
INSTI resistance among incident HIV infections | 24 months
  The % of incident maternal and infant HIV infections found to have INSTI resistance
Inadequate infant growth | 24 months
  The % of infants with Z-score >=2SD below WHO norms for length-for-age or weight-for-age
Infant microcephaly | 24 months
  Infants with head circumference >=2SD below WHO norms for head-circumference for age

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Zash, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States
- Botswana Harvard AIDS Institute Partnership, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: Yes
Researchers who provide a methodologically sound proposal (approved by the Tshireletso study team) for use of the data, including for pooling of data on the safety of medications in pregnancy and lactation to achieve aims, that have ethics approval from all involved institutions. Researchers of approved proposals will need to sign a Data Use Agreement with BIDMC before receiving the data.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available starting 3 months after the publication of the main outcomes of the Tshireletso study and be available until the end of the funding period for this study.